CLINICAL TRIAL: NCT00757276
Title: Copeptin in the Diagnosis and Differential Diagnosis of Diabetes Insipidus. The CoSIP-Study
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: EKBB 68/08
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Diabetes Insipidus
Keywords: Copeptin; Diabetes insipidus; diagnostic marker; Vasopressin; antidiuretic hormone (ADH)
MeSH Terms: conditions — Diabetes Insipidus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — bood sampling

GROUPS / COHORTS (1):
- 1: All patients > 18 years who are tested for the diagnosis of DI because of a history of polyuria (> 40 ml/kg per 24 hours) in the presence of polydipsia Patients with known DI will be contacted whether they agree to participate in the study and to undergo again a water deprivation test to measure copeptin to confirm the diagnosis.
  The investigators hypothesize that basal copeptin levels can reliably differentiate between the 5 groups(central, nephrogenic, psychogenic and partial forms) with a sensitivity and specificity >80%.

SUMMARY:
Evaluation of Copeptin in the differential diagnosis of diabetes insipidus.

DETAILED DESCRIPTION:
Background:

Plasma arginine vasopressin (AVP) measurement is recommended for the differential diagnosis of diabetes insipidus and polydipsia. However, AVP measurement is cumbersome. AVP is derived from a larger precursor peptide along with copeptin, which is a more stable peptide directly mirroring the production of AVP. Copeptin can be assayed readily in plasma.

Aim: To evaluate the diagnostic accuracy of copeptin levels in the diagnosis and differential diagnosis of diabetes insipidus.

Design: Prospective, observational multicenter study.

Setting: Department of Endocrinology, University Hospital of Basel

Patients: Patients with suspected or known central (complete or partial), nephrogenic (complete or partial) or psychogenic diabetes insipidus undergoing a standardized water deprivation test.

Intervention: All patients with suspected or known diabetes insipidus will undergo an overnight water deprivation test and a standardized water deprivation test, as routinely performed in the diagnostic evaluation of diabetes insipidus. Plasma AVP and copeptin will be measured at baseline (8 am before start of thirsting), and hourly during the water deprivation test.

Study hypothesis: Copeptin levels will provide a better diagnostic accuracy in the diagnosis and differential diagnosis of diabetes insipidus as compared to AVP measurement.

Analysis: We will study 5 groups of patients: A) Patients with complete central diabetes insipidus, B) Patients with partial central diabetes insipidus, C) Patients with complete nephrogenic diabetes insipidus, D) Patients with partial nephrogenic diabetes insipidus and E) Patients with psychogenic diabetes insipidus. All groups will consist of 10 patients based on the following assumptions: Based on pilot studies we assume that patients in group A) will have copeptin values of 2.5 ± 1.0; Group B) 3.0 ± 1.0, Group C) 15.0 ± 5; Group D) 6 ± 2.0 and Group E) 4.0 ± 1.0 pmol/L. This results in a power of 90% to detect a difference in copeptin levels of 0.8pmol/L between the closest two groups, i.e. patients with partial central Diabetes insipidus and patients with psychogenic Diabetes insipidus.

Significance: The measurement of copeptin will allow a better discrimination of patients with diabetes insipidus, especially for the discrimination of partial central and nephrogenic and psychogenic diabetes insipidus.

ELIGIBILITY:
Inclusion Criteria:

* All patients > 18 years who are tested for the diagnosis of DI because of a history of polyuria (> 40 ml/kg per 24 hours) in the presence of polydipsia Patients with known DI will be contacted whether they agree to participate in the study and to undergo again a water deprivation test to measure copeptin to confirm the diagnosis.

Exclusion Criteria:

* Polyuria of other origin, i.e. prostate hyperplasia, diabetes mellitus.
* Pregnancy
* The investigators do not perform the water deprivation test in patients with: *renal insufficiency

  * uncontrolled diabetes mellitus
  * hypovolemia of any cause
  * uncorrected deficiency of adrenal or thyroid hormones
* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients >18 years who are tested for the diagnosis of DI because of a history of polyuria (>40ml/kg per 24 hours) in the presence of polydipsia Patients with known DI will be contacted whether they agree to participate in the study and to undergo again a water deprivation test to measure copeptin to confirm the diagnosis.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Diagnosis of diabetes insipidus(DI) centralis versus psychogenic DI | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, Prof. Dr. med., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Basel, Switzerland

REFERENCES:
- [Derived] Atila C, Winzeler B, Chifu I, Fassnacht M, Refardt J, Christ-Crain M. A post-hoc internal validation of arginine-stimulated copeptin cut-offs for diagnosing AVP deficiency (central diabetes insipidus). Pituitary. 2025 Apr 26;28(3):53. doi: 10.1007/s11102-025-01523-2. PMID 40281371
- [Derived] Ebrahimi F, Urwyler SA, Betz MJ, Christ ER, Schuetz P, Mueller B, Donath MY, Christ-Crain M. Effects of interleukin-1 antagonism and corticosteroids on fibroblast growth factor-21 in patients with metabolic syndrome. Sci Rep. 2021 Apr 12;11(1):7911. doi: 10.1038/s41598-021-87207-w. PMID 33846498
- [Derived] Bologna K, Cesana-Nigro N, Refardt J, Imber C, Vogt DR, Christ-Crain M, Winzeler B. Effect of Arginine on the Hypothalamic-Pituitary-Adrenal Axis in Individuals With and Without Vasopressin Deficiency. J Clin Endocrinol Metab. 2020 Jul 1;105(7):dgaa157. doi: 10.1210/clinem/dgaa157. PMID 32236441
- [Derived] Winzeler B, Cesana-Nigro N, Refardt J, Vogt DR, Imber C, Morin B, Popovic M, Steinmetz M, Sailer CO, Szinnai G, Chifu I, Fassnacht M, Christ-Crain M. Arginine-stimulated copeptin measurements in the differential diagnosis of diabetes insipidus: a prospective diagnostic study. Lancet. 2019 Aug 17;394(10198):587-595. doi: 10.1016/S0140-6736(19)31255-3. Epub 2019 Jul 11. PMID 31303316
- [Derived] Urwyler SA, Timper K, Fenske W, de Mota N, Blanchard A, Kuhn F, Frech N, Arici B, Rutishauser J, Kopp P, Stettler C, Muller B, Katan M, Llorens-Cortes C, Christ-Crain M. Plasma Apelin Concentrations in Patients With Polyuria-Polydipsia Syndrome. J Clin Endocrinol Metab. 2016 May;101(5):1917-23. doi: 10.1210/jc.2016-1158. Epub 2016 Mar 11. PMID 26967692
- [Derived] Timper K, Fenske W, Kuhn F, Frech N, Arici B, Rutishauser J, Kopp P, Allolio B, Stettler C, Muller B, Katan M, Christ-Crain M. Diagnostic Accuracy of Copeptin in the Differential Diagnosis of the Polyuria-polydipsia Syndrome: A Prospective Multicenter Study. J Clin Endocrinol Metab. 2015 Jun;100(6):2268-74. doi: 10.1210/jc.2014-4507. Epub 2015 Mar 13. PMID 25768671